CLINICAL TRIAL: NCT04941040
Title: Hemodynamic Effects of Opioid Free Anesthesia Versus Opioid Anesthesia on Adult Patients Undergoing Craniotomies for Supratentorial Tumors. Randomized Controlled Trial
Brief Title: Opioid Free VS Opioid Anesthesia for Craniotomies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Rania Samir Fahmy, Assistant professor of Anesthesia, ICU and pain medicine, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: N 56-2016/MD
Record Dates: First submitted 2021-06-12; First posted 2021-06-28 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Supratentorial Neoplasms
Keywords: Opioid free Anesthesia; Craniotomies; Dexmedetomidine; Ketamine; Fentanyl; Lidocaine; Magnesium sulphate; supratentorial tumors
MeSH Terms: conditions — Supratentorial Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid free anesthesia (Experimental): patients are going to receive intraoperative analgesics other than opioids
  Interventions: Drug: Opioid free anesthetics
- Opioid anesthesia (Active Comparator): patients are going to receive intraoperative opioid analgesics
  Interventions: Drug: Opioid Anesthetics

INTERVENTIONS:
Drug: Opioid free anesthetics — Patients will receive over the 10 minutes prior to induction:
  * Acetaminophen 1 gm i.v. infusion in 100ml over 10 minutes.
  * Ketorolac 30 mg i.v. infusion in100 ml over 10 minutes.
  * Mg SO4 loading dose 30 mg/kg i.v. infusion in 100 ml over 10 minutes.
  * Dexmedetomidine loading dose 1 μg/kg i.v. infusion.
  * Lidocaine loading dose 1.5 mg/kg i.v. infusion.
  * Ketamine loading dose 0.25 mg/kg i.v. infusion.
  The weight based doses of dexmedetomidine, lidocaine, ketamine will be prepared on 20 ml syringe and infused over 10 minutes prior to induction. In a dose of 0.1 ml/kg
  Then after induction maintenance analgesic infusion will start in a rate that ranges from 0.025 to 0.05 ml/kg/h which is equivalent to:
  * Dexmedetomidine 0.25-0.5 μg/kg/h
  * Lidocaine 0.375-0.75 mg/kg/h
  * Ketamine 0.0625- 0.125 mg/kg/h
  Other Names: OFA
  Arms: Opioid free anesthesia
Drug: Opioid Anesthetics — Placebo equivalent to acetaminophen, ketorolac, magnesium sulphate will be infused as 100 ml normal saline each over 10 minutes ,patients will receive fentanyl 2 μg/kg loading dose which will be prepared over 20 ml syringe and infused over 10 minutes prior to induction, Then after induction maintenance of analgesic infusion by fentanyl 0.5-1 μg/kg/h.
  Other Names: OA
  Arms: Opioid anesthesia

SUMMARY:
Hemodynamic control during craniotomies can be a bit hectic specially during periods of intense noxious stimulation. For long anesthesiologists used high doses of opioids such as fentanyl and remifentanyl to provide analgesia with a good hemodynamic control during intraoperative period in patients undergoing craniotomies. However, the use of opioids was not devoid of side effects. Exploring other anesthetic plans using multiple opioid free anesthetic adjuvants that have analgesic effects given together in small doses appear to be appealing plan. This idea is the basis of our proposed study in which we compare the hemodynamic effects of using opioid free anesthesia versus opioid anesthesia in cranial surgeries.

DETAILED DESCRIPTION:
Anesthesia for craniotomies can be very challenging because of the presence of periods of noxious stimuli that interposes with periods of little stimulation which makes hemodynamic control a little bit more complicated. Intraoperative episodes of hypertension during periods of intense stimulations and early postoperative hypertension may lead to serious complications as post craniotomy intracranial hemorrhage and vasogenic brain edema. Anesthetic techniques based on usage of high doses of potent opioid analgesics such as fentanyl and remifentanil have been widely popular among anesthesiologists. However, the intra operative use of large bolus doses or continuous infusions of potent opioids may be associated with postoperative hyperalgesia and increased analgesic consumption.

More recently, concerns have arisen about impaired healing,immunosuppression,and worsening of oncologic outcomes with systemic opioids. Another technique that started gaining its popularity is opioid free anesthesia (OFA) technique whose corner stone is depending on multiple anesthetic adjuvants that have analgesic effects, , therefore when given together in small doses they result in good anesthesia with less side effects and faster recovery compared with opioids. This technique has been successfully used in anesthesia for bariatric surgeries combining multiple drugs as dexmedetomidine, lidocaine, ketamine, ketorolac and magnesium.

Dexmedetomidine is a highly selective α2-adrenoceptor agonist with sedative, anxiolytic and analgesic properties that has minimal effects on respiratory drive. Although preoperative intravenous dexmedetomidine administration is associated with a reduction in postoperative pain intensity, analgesic consumption and nausea, the analgesic property of dexmedetomidine is less effective compared with opioids. Intravenous lidocaine has been described as having analgesic, anti-hyperalgesic, and anti-inflammatory properties. Intravenous lidocaine infusion in the perioperative period is safe and has clear advantages, such as decreased intra operative anesthetic requirements, lower pain scores, reduced postoperative analgesic requirements, as well as faster recovery. In addition to ketamine magnesium is also reported to enhance analgesia by blocking NMDA receptor, also magnesium has the properties of a sympatholytic and has been introduced as a safe component of balanced anesthesia.

This comparative study between Opioid free anesthesia (OFA) and Opioid anesthesia (OA) aims to compare the effect of both techniques on intra operative hemodynamics, intracranial tension and recovery in cranial surgeries for supratentorial tumors.

After obtaining an informed written consent from the patients or their responsible relative, patients will be divided into 2 groups randomly using computer software (research randomizer.org); Opioid free Anesthesia group (OFA) and Opioid Anesthesia group (OA). To assure blindness, numbers will be concealed by closed envelope, analgesic infusions will prepared by a clinical pharmacist not included in data collection and the attending anesthetist will be blinded to the type of analgesic solution injected.

Over 10 minutes prior to induction of analgesia patients in the OFA group will receive small doses of demedetomidine, ketamine, lidocaine and magnesium along with ketorlac and acetaminophen. an infusion afterwards will be administered through the operation containing dexmedetomidine, ketamine and lidocaine. In the OA group, over 10 minutes, patients will receive a loading dose of fentanyl followed by fentanyl infusion through the operation. General anesthesia will be induced using the same drugs and the same parameters in both groups after the completion of the initial analgesic infusions The primary outcome parameter will be the percentage of patients experiencing hemodynamic instability at Burr Hole (defined as recording an increase or decrease of the mean arterial blood pressure by 25 % of the baseline reading) Assuming the rate of hemodynamic instability (defined as increase or decrease of the mean blood pressure by 25 % of the baseline reading) would be 40 % in the control arm, a clinically meaningful reduction of the rate of hemodynamic instability to 10 % in the investigational arm with a statistical power of 80 % and an alpha error of less than 0.05 would require recruiting 29 patients in each group (a total of 58 patients).

Continuous data will be presented as mean + (SD). Categorical variables will be represented as frequencies and percentages. According to the type of data Comparison between the two groups will be performed using either Chi square test or Fisher's exact test. Hemodynamic variables will be compared to baseline using repeated measures analysis of variance (ANOVA) with post hoc scheffe's test for positive data. P values less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* ASA Ι and II.
* Patients undergoing surgeries for removal of supratentorial tumors.
* Age (18-60) years.
* Both sexes.

Exclusion Criteria:

* Impaired renal functions.
* Systemic hypertension.
* Dysrhythmia.
* Heart failure.
* Glasgow coma scale less than 12.
* The need for postoperative ventilation.
* History of allergy to the study drugs.
* Surgeries lasting more than 6 hours.
* Pregnancy.
* Bronchial asthma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2021-10-03 (Actual); Study Completion 2021-10-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients experiencing a change in mean arterial pressure at time of Burr Hole | During Burr hole surgery
  Defined as recording an increase or decrease of the mean arterial blood pressure by more than 25 % from baseline readings at the time of burr hole

SECONDARY OUTCOMES:
HR (heart rate) in beats/min | Baseline, pre-induction, pre-intubation, after intubation, skin incision, burr hole, dural incision, dural closure, skin closure, every 30 minutes intraoperative till extubation, time of extubation, every 15 minutes for 2 hours in PACU.
  Hemodynamic parameter recorded during the study
Brain relaxation score | At the time of dural incision
  Defined as 1= excellently relaxed, 2= satisfactory relaxed, 3= leveled, 4=bulging
Number of patients requiring antihypertensive medication | Throughout the operation
  Number of patients needing nitroglycerine infusion in each group was recorded together with total amount infused
Number of patients requiring medication to increase blood pressure | Throughout the operation
  Number of patients needing ephedrine in each group was recorded together with total amount infused.
Time to extubation | At the end of the operation, the time from the discontinuation of inhalation agents till extubation
  Defined as the time between the discontinuation of inhalation agents and extubation
Ramsay Sedation Scale (RSS) | every 30 minutes for 2 hours postoperative
  to assess the postoperative sedation, it is a scale from 1 to 6. It provides three levels of 'awake' states (score 1-3) and three levels of 'asleep' states (score 4-6). A score of 2 (patient is cooperative, orientated and tranquil)
Systolic blood pressure (SBP) in mmhg | Baseline, pre-induction, pre-intubation, after intubation, skin incision, burr hole, dural incision, dural closure, skin closure, every 30 minutes intraoperative till extubation, time of extubation, every 15 minutes for 2 hours in PACU.
  Hemodynamic parameter recorded during the study
Mean arterial blood pressure (MAP) in mmhg | Baseline, pre-induction, pre-intubation, after intubation, skin incision, burr hole, dural incision, dural closure, skin closure, every 30 minutes intraoperative till extubation, time of extubation, every 15 minutes for 2 hours in PACU.
  Hemodynamic parameter recorded during the study

CONTACTS AND LOCATIONS:
Overall Officials: Rania S Fahmy, Principal Investigator — Kasr Al Ainy, Faculty of medicine, Cairo university
Locations (1):
- Kasr El Aini Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uyar AS, Yagmurdur H, Fidan Y, Topkaya C, Basar H. Dexmedetomidine attenuates the hemodynamic and neuroendocrinal responses to skull-pin head-holder application during craniotomy. J Neurosurg Anesthesiol. 2008 Jul;20(3):174-9. doi: 10.1097/ANA.0b013e318177e5eb. PMID 18580347
- [Background] Basali A, Mascha EJ, Kalfas I, Schubert A. Relation between perioperative hypertension and intracranial hemorrhage after craniotomy. Anesthesiology. 2000 Jul;93(1):48-54. doi: 10.1097/00000542-200007000-00012. PMID 10861145
- [Background] Angst MS, Clark JD. Opioid-induced hyperalgesia: a qualitative systematic review. Anesthesiology. 2006 Mar;104(3):570-87. doi: 10.1097/00000542-200603000-00025. PMID 16508405
- [Background] Mulier JP. Perioperative opioids aggravate obstructive breathing in sleep apnea syndrome: mechanisms and alternative anesthesia strategies. Curr Opin Anaesthesiol. 2016 Feb;29(1):129-33. doi: 10.1097/ACO.0000000000000281. PMID 26595546
- [Background] Cortinez LI, Hsu YW, Sum-Ping ST, Young C, Keifer JC, Macleod D, Robertson KM, Wright DR, Moretti EW, Somma J. Dexmedetomidine pharmacodynamics: Part II: Crossover comparison of the analgesic effect of dexmedetomidine and remifentanil in healthy volunteers. Anesthesiology. 2004 Nov;101(5):1077-83. doi: 10.1097/00000542-200411000-00006. PMID 15505442
- [Background] Lauwick S, Kim DJ, Michelagnoli G, Mistraletti G, Feldman L, Fried G, Carli F. Intraoperative infusion of lidocaine reduces postoperative fentanyl requirements in patients undergoing laparoscopic cholecystectomy. Can J Anaesth. 2008 Nov;55(11):754-60. doi: 10.1007/BF03016348. PMID 19138915
- [Background] Syeda S, Palaniswamy SR, Sriganesh K. Opioid Free Analgesia With Dexmedetomidine for Craniotomy in an Obese Patient With Obstructive Sleep Apnea and Difficult Airway. Asian J Anesthesiol. 2020 Jun 1;58(2):76-77. doi: 10.6859/aja.202006_58(2).0007. Epub 2020 Jul 24. No abstract available. PMID 33171574